CLINICAL TRIAL: NCT04106141
Title: Effect of Changing the Activation Frequency of the Arch Wires on the Rate of Leveling and Alignment in Moderate Crowding Cases
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Seif-Allah Ahmed Sherif Nasr, masters student, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ORTH 3-3-4
Record Dates: First submitted 2019-09-23; First posted 2019-09-26 (Actual); Last update posted 2019-09-26 (Actual); Status verified 2019-09

CONDITIONS: Leveling and Alignment of Teeth

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (Other)
  Interventions: Other: 4 weeks changing of archwire
- intervention group (Active Comparator)
  Interventions: Other: 6 weeks changing of archwire

INTERVENTIONS:
Other: 6 weeks changing of archwire — changing the archwire after 6 weeks instead of 4 weeks
  Arms: intervention group
Other: 4 weeks changing of archwire — changing the archwire every 4 weeks
  Arms: control group

SUMMARY:
Leveling and alignment is the first stage in the orthodontic treatment, performed for every patient .The archwire are usually changed every 4 weeks for reactivation of the force on the teeth. However, this means that large number of appointments and archwires are required. On the other hand, there is a lack of evidence that less number of appointments with longer time intervals between the visits and less number of wires will give the same effect.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients aged (18~33)
* CVMI = 6
* Moderate crowding (4-8) as described by Laura mitchel
* No extractions required

Exclusion Criteria:

* Growing patients
* Previous orthodontic treatment
* Missing teeth other than the wisdoms

Ages: 18 Years to 33 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 22 (Estimated)
Dates: Start 2020-01-01 (Estimated); Primary Completion 2021-09-04 (Estimated); Study Completion 2021-11-09 (Estimated)

PRIMARY OUTCOMES:
Degree of alignment of teeth | 5 months
  the teeth are aligned together by using Little irregularity index to measure the decrease in the discrepency in each digital model taken after changing of the wire